CLINICAL TRIAL: NCT06627972
Title: Is THERE a RELATIONSHIP BETWEEN PERIODONTAL CONDITION and ASPROSIN LEVEL in GINGIVAL CREVICULAR FLUID?
Brief Title: Asprosin Level in Individuals with Periodontal Disease
Acronym: ALIGCF
Status: Completed | Type: Observational
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Osman Fatih Arpag, Principal investigator, Mustafa Kemal University
Other Study IDs: DHFDUP/2022-0002
Record Dates: First submitted 2024-10-01; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Periodontitis; Periodontal Health; Gingivitis
Keywords: gingival crevicular fluid; asprosin hormone; periodontal diseases; tumour necrosis factor alpha
MeSH Terms: conditions — Periodontitis; Gingivitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- periodontal health group: Periodontal parameters were recorded at first visit and the fluid samples were collected from participants.
- Gingivitis group: Periodontal parameters were recorded at first visit and the fluid samples were collected from participants.
- periodontitis group: Periodontal parameters were recorded at first visit and the fluid samples were collected from participants.

SUMMARY:
The aim of this study was to investigate the levels of asprosin hormone and tumour necrosis factor alpha (TNF-α) in gingival crevicular fluids and to compare its level with those in saliva and serum in patients with gingivitis and periodontitis.

DETAILED DESCRIPTION:
This study is investigating the level of asprosin hormone in gingival crevicular fluid of patients with periodontal diseases such as gingivitis and periodontitis, and observing the healthy patient in terms of the hormone levels, as well. 75 volunteer patients aged 18-45 years old were included in this study. These patients were divided equally to three groups: Group I; periodontal health, Group II; gingivitis, Group III; periodontitis.The body fluids including serum, saliva and gingival crevicular fluid were collected from this participants according to the proper protocol and their storage was provided under certain conditions. ELISA tests for asprosin and Tumour necrosis factor alpha were made in laboratory. Also, clinical measurements such as plaque index, bleeding on probing, probing pocket depth were recorded at first visit day of the participants. The data were analysed according to the different periodontal conditions, and correlated with asprosin hormone and tumour necrosis factor alpha level in gingival crevicular fluid, serum and saliva.

ELIGIBILITY:
Exclusion Criteria:

* Those with any systemic disease
* Individuals who take medication regularly
* Pregnant or lactating women
* Individuals with menopause and anthropause
* Those who have undergone any periodontal treatment in the last six months
* Smokers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants who applied to the Periodontology Department in Adiyaman University, Faculty of Dentistry were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Asprosin level | Day 1
  Asprosin level (ng/mL) in gingival crevicular fluid, serum and saliva.

SECONDARY OUTCOMES:
TNF-alpha levels | Day 1
  TNF-alpha level (pg/mL) in gingival crevicular fluid, serum and saliva
Plaque index | Day 1
  The index was recorded from all participants as numerical between 0-3
bleeding on probing | Day 1
  The bleeding on probing is stated by percentage. the ratio of the number of sites with bleeding gingiva on probing around teeth to total surfaces of all examined teeth
probing pocket depth | Day 1
  The parameters were recorded as mm in all participant. The probing pocket depth is measured from the marginal gingiva to bottom of pocket using a periodontal probe, from six surfaces of each tooth.
body mass index | Day 1
  the weight and height is combined to report BMI in kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Abdulsamet Tanık, PhD, Study Chair — Adiyaman University
Locations (1):
- Adiyaman University, Faculty of Dentistry, Adıyaman, Turkey (Türkiye)

REFERENCES:
- [Background] Shojaee M, Fereydooni Golpasha M, Maliji G, Bijani A, Aghajanpour Mir SM, Mousavi Kani SN. C - reactive protein levels in patients with periodontal disease and normal subjects. Int J Mol Cell Med. 2013 Summer;2(3):151-5. PMID 24551806
- [Background] Gul SNS, Eminoglu DO, Laloglu E, Aydin T, Dilsiz A. Salivary and serum asprosin hormone levels in the 2018 EFP/AAP classification of periodontitis stages and body mass index status: a case-control study. Clin Oral Investig. 2024 Jan 13;28(1):91. doi: 10.1007/s00784-024-05494-9. PMID 38217801
- [Background] de Molon RS, Rossa C Jr, Thurlings RM, Cirelli JA, Koenders MI. Linkage of Periodontitis and Rheumatoid Arthritis: Current Evidence and Potential Biological Interactions. Int J Mol Sci. 2019 Sep 13;20(18):4541. doi: 10.3390/ijms20184541. PMID 31540277
- [Background] Afacan B, Ozturk VO, Pasali C, Bozkurt E, Kose T, Emingil G. Gingival crevicular fluid and salivary HIF-1alpha, VEGF, and TNF-alpha levels in periodontal health and disease. J Periodontol. 2019 Jul;90(7):788-797. doi: 10.1002/JPER.18-0412. Epub 2018 Dec 11. PMID 30536725
- [Derived] Tutus S, Tanik A, Arpag OF, Onderci M. Is there a relationship between periodontal conditions and asprosin levels in gingival crevicular fluid, saliva and serum? BMC Oral Health. 2025 Apr 29;25(1):651. doi: 10.1186/s12903-025-06014-1. PMID 40301876